CLINICAL TRIAL: NCT03804450
Title: Magnetic Resonance Imaging Assessment of Pulp Regeneration Following Regenerative Endodontic Procedures in Mature Teeth
Brief Title: Magnetic Resonance Imaging (MRI) of Pulp Regeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Noha Mohamed El Kateb, Assistant lecturer, Faculty of dentistry, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15012017
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pulp Necroses; Periapical Lesion; Regeneration
Keywords: Mature teeth; Necrotic teeth; REPs; Biodentine; MRI; CBCT
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The root canals were instrumented using Pro-taper next rotary files till size X3. REPs via blood clot using calcium hydroxide were then applied
  Interventions: Procedure: Regenerative endodontic procedures (REPs)
- Control group (Experimental): The root canals were instrumented using Pro-taper next rotary files till size X5. REPs via blood clot using calcium hydroxide were then applied.
  Interventions: Procedure: Regenerative endodontic procedures (REPs)

INTERVENTIONS:
Procedure: Regenerative endodontic procedures (REPs) — Instrumentation using rotary Pro-Taper Next, disinfection using sodium hypochlorite and calcium hydroxide as intracanal medication followed by induction of blood and application of Biodentine as a cervical plug.
  Other Names: Pulp Regeneration

SUMMARY:
The present study was conducted to test whether pulp-like tissue can be regenerated in mature teeth with closed apex? And whether the size of the apical diameter affects the success of REPs? And whether Magnetic resonance imaging (MRI) can be used to quantitatively assess the vitality of the regenerated pulp-like tissue.

DETAILED DESCRIPTION:
Regenerative endodontic procedures via blood clot were done on 18 mature anterior necrotic teeth with periapical lesions. The teeth were randomly assigned into two groups according to the size of the apical diameter of the rotary files used for instrumentation.

In the test group, rotary instrumentation was done using Pro-taper Next till size X3, while in the control group, instrumentation was done till size X5.

Calcium hydroxide was used as an intracanal medication for 1-2 weeks. Calcium hydroxide was then washed away using 1.5%NaOCl, followed by induction of blood using pre-curved K-fi;e #25 2mm past the radiographic apex. Biodentine was then used as a cervical plug over the blood clot followed by resin-modified glass ionomer cement and composite resin as coronal restoration.

MRI was used to assess the vitality of the regenerated pulp-like tissue, where the signal intensity of the regenerated pulp-like tissue was measured after 3,6 and 12 months follow up and compared to the normal contralateral teeth. In addition, sensibility tests using cold test and electric pulp testing were used to assess vitality of regenerated pulp-like tissue after 3,6,9 and 12 months. Cone beam computed tomography (CBCT) was also used to assess the healing of the periapical lesion after 12 months.

ELIGIBILITY:
Inclusion Criteria

* Upper anterior mature teeth with single canals.
* Necrotic teeth
* Presence of periapical lesion.

Exclusion Criteria:

* Presence of systemic diseases.
* Presence of stainless steel wires o brackets
* Vital immature teeth with open apex

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
MRI assessment of pulp-like tissue regeneration | 12 months
  Signal intensity of the regenerated pulp-like tissue was quantitatively measured in both test and control groups after 3,6 and 12 months follow up and compared to the contralateral normal teeth.

SECONDARY OUTCOMES:
Healing of the periapical lesion | 12 months
  Cone beam computed tomography (CBCT) was used to assess the healing of the periapical lesion after 12 months follow up period.
Positive pulpal response | 12 months
  The positive response to sensibility tests using cold test and electric pulp tester was done after 3,6,9 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] El-Kateb NM, Abdallah AM, ElBackly RN. Correlation between pulp sensibility and magnetic resonance signal intensity following regenerative endodontic procedures in mature necrotic teeth- a retrospective cohort study. BMC Oral Health. 2024 Mar 13;24(1):330. doi: 10.1186/s12903-024-04095-y. PMID 38481211